CLINICAL TRIAL: NCT04314375
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Budesonide Extended-release Tablets n Pediatric Subjects Aged 5 to 17 Years With Active, Mild to Moderate Ulcerative Colitis
Brief Title: Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Budesonide Extended-release Tablets in Pediatric Subjects Aged 5 to 17 Years With Active, Mild to Moderate Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUUC4991
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose Budesonide (Experimental)
  Interventions: Drug: Low Dose Budesonide
- High Dose Budesonide (Experimental)
  Interventions: Drug: High Dose Budesonide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Budesonide — 3 milligrams once daily for ages 5 to 11 years 11 months. 6 milligrams once daily for ages 12 to 17 years.
  Arms: Low Dose Budesonide
Drug: High Dose Budesonide — 6 milligrams once daily for ages 5 to 11 years 11 months. 9 milligrams once daily for ages 12 to 17 years.
  Arms: High Dose Budesonide
Drug: Placebo — Matching placebo once daily.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, study to evaluate the efficacy, safety, and pharmacokinetics (PK) of budesonide extended-release tablets for the induction of remission in pediatric subjects, with active, mild to moderate ulcerative colitis (UC). Subjects will be permitted to continue taking background oral or rectal 5-aminosalicylate (5-ASA) products.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of UC is based on:

  * Clinical history
  * Characteristic endoscopic findings
  * Histopathology results from biopsies
* Age 5 to 17 years, inclusive, at Screening. Subjects should weigh greater than 13.6 kg at Baseline.
* Active UC of mild or moderate severity, defined as a total Mayo score between 4 and 10, inclusive, with rectal bleeding subscore of ≥ 1, stool frequency subscore of ≥1 and an endoscopy subscore of ≥ 1.
* If on a background oral or rectal 5-ASA, the dose and formulation have remained unchanged for at least 6 weeks prior to Visit 2 (randomization), Baseline and the subject is willing to remain on the same formulation and dose for the duration of the study.

Exclusion Criteria:

1. Current or prior diagnosis of Crohn's disease or indeterminate colitis.
2. Limited distal proctitis (disease involving only the first 15 centimeters or less proximal to the anal verge.
3. Severe UC, defined as total Mayo score >10.
4. Not currently in an active phase or flare, defined as a total Mayo score <4, or Mayo score between 4 and 10, but Mayo subscore of 0 for rectal bleeding, stool frequency or endoscopy.
5. Infectious colitis (based on positive microbiologic tests at Screening) or any recent history of infectious colitis (within 30 days prior to Screening).
6. Prior gastrointestinal surgery, except appendectomy or hernia (e.g., inguinal, umbilical).

   NOTE: Prior cholecystectomy is not exclusionary if more than 1 year prior to Screening.
7. Evidence or history of toxic megacolon or bowel resection.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of subjects who achieve clinical remission at Day 56, defined as a total Mayo score of ≤ 1 with subscores of 0 for both rectal bleeding and stool frequency, and a subscore of ≤ 1 for endoscopy. | 56 days
  The primary efficacy endpoint is the proportion of subjects who achieve clinical remission at Day 56, defined as a total Mayo score of ≤ 1 with subscores of 0 for both rectal bleeding and stool frequency, and a subscore of ≤ 1 for endoscopy. The Mayo score is a composite index score based on 4 components: stool frequency (subject reported), rectal bleeding (subject reported), findings of endoscopy, and the physician's rating of disease activity. Each component is scored from 0 to 3, with total scores range from 0 to 12 with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Proportion of subjects who achieve a Mayo rectal bleeding subscale score of 0 at Day 56. | 56 days
  Proportion of subjects who achieve a Mayo rectal bleeding subscale score of 0 at Day 56. The Mayo score is a composite index score based on 4 components: stool frequency (subject reported), rectal bleeding (subject reported), findings of endoscopy, and the physician's rating of disease activity. Each component is scored from 0 to 3, with total scores range from 0 to 12 with higher scores indicating more severe disease.
Proportion of subjects who achieve a Mayo stool frequency subscale score of 0 at Day 56. | 56 days
  Proportion of subjects who achieve a Mayo stool frequency subscale score of 0 at Day 56. The Mayo score is a composite index score based on 4 components: stool frequency (subject reported), rectal bleeding (subject reported), findings of endoscopy, and the physician's rating of disease activity. Each component is scored from 0 to 3, with total scores range from 0 to 12 with higher scores indicating more severe disease.
Proportion of subjects who achieve a Mayo endoscopy subscale score of 0 or 1 at Day 56. | 56 days
  Proportion of subjects who achieve a Mayo endoscopy subscale score of 0 or 1 at Day 56. The Mayo score is a composite index score based on 4 components: stool frequency (subject reported), rectal bleeding (subject reported), findings of endoscopy, and the physician's rating of disease activity. Each component is scored from 0 to 3, with total scores range from 0 to 12 with higher scores indicating more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (4):
- United States (4):
  - Bausch Health Site 008, Garden Grove, California
  - Bausch Health Site 003, Indianapolis, Indiana
  - Bausch Health Site 006, The Bronx, New York
  - Bausch Health Site 010, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided